CLINICAL TRIAL: NCT05593172
Title: Different Courses of Change in Connectivity After mTBI Depending on Cognitive Reserve and How This is Related to Symptoms and Symptom Resolution?
Brief Title: Change in Connectivity After mTBI Depending on Cognitive Reserve
Status: Completed | Type: Observational
Sponsor: Danderyd Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: fMRICogRev
Record Dates: First submitted 2022-10-10; First posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Mild Traumatic Brain Injury
Keywords: rs-fMRI; Cognitive reserve; Fatigue; Visual disturbances
MeSH Terms: conditions — Brain Concussion; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mild traumatic brain injury: 15 consecutive patients presenting at the emergency departement with mild traumatic brain injury
- Minor orthopedic injury: 15 patients, recruited during the same time-frame as the mTBI-patients, presenting at the emergency departement with a minor orthopedic injury

SUMMARY:
The purpose of this study is to investigate the role of cognitive reserve in change in connectivity in the brain (measured with functional magnetic resonance imaging, fMRI) and how this is related to symptoms and symptom resolution.

DETAILED DESCRIPTION:
The population-based rate of mild traumatic brain injury (mTBI) is estimated to exceed 600/100000 population per year in total, if including only patients seeking emergency care the estimated rate is approximately 100-300/100000. Many patients recover within 3 months after injury but a sustainable proportion suffer from persisting symptoms, for instance fatigue, headaches, irritability. As conventional neuroimaging techniques have failed to detect the subtle alterations that may be important for prognosis and long-term outcome after mTBI, studies using fMRI have shown some interesting results. Other variables, for instance demographic and cognitive variables, also need to be incorporated with imaging biomarkers when investigating the relationship between fMRI biomarkers with outcome after mTBI. A marker related to demographic status and cognition that have shown to be relevant for outcome in brain injury or pathology is cognitive reserve. Cognitive reserve is defined as an aspect of the brain's function or structure that impacts the relationship between injury/pathology and outcome. Higher cognitive reserve is related to better outcome in conditions ranging from Alzheimer, MS and mTBI.

In this study 15 patients with mTBI and 15 patients with minor orthopedic injury underwent assessment, including cognitive testing, self-assessment of symptoms, testing of visual functions and resting-state fMRI at approximately one week after injury and 4 months after injury. Cognitive reserve was assessed with a lexical decision test designed to measure pre-morbid IQ.

Descriptive statistics will be used to depict demographics, injury characteristics, results on neuropsychological tests and psychological screening instruments. Multi-subject and multi-session analysis based on general linear model will be performed and assessed using statistical tools including regression analysis and 2-way ANOVA.

ELIGIBILITY:
Inclusion Criteria mTBI group:

* presenting at the emergency departement between January 2015 and April 2016 due to an mTBI to such an extent that CT was indicated.
* mTBI was defined by a Glasgow Coma Scale score between 13-15 and one or more of the following symptoms: <30 minutes loss of consciousness, <24 hours post-traumatic amnesia and/or a transient neurological deficit according to the WHO Collaborating center of Neurotrauma Task Force

Inclusion Criteria orthopedic group:

* presenting at the emergency departement between January 2015 and April 2016 due to minor traumatic injuries to the hand, foot, arm or leg that did not require surgical intervention.

Exclusion Criteria:

* uncertain duration of loss of consciousness
* contraindications to MR
* previously acquired brain injury, a progressive neurological disorder or another injury/illness with short expected survival
* were dependent of help in daily living before the current damage
* severe visual impairment
* non-Swedish speaking.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants were all adults presenting at the emergency departement at Danderyd Hospital, (Stockholm, Sweden) during the given time frame, with minor head injury or minor orthopedic injury. An upper age limit of 40 years were set due to avoiding interference with age-related visual disturbances.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-01-24 (Actual); Primary Completion 2016-05-03 (Actual); Study Completion 2016-05-03 (Actual)

PRIMARY OUTCOMES:
State fatigability | Measured at approximately one week after injury
  Difference between score during the first 60 and the last 60 seconds of the Digit Symbol Substitution Test/Coding (DSST). The lower the score, the stronger the indication of fatigability
State fatigability | Measured at approximately 4 months after injury
  Difference between score during the first 60 and the last 60 seconds of the Digit Symbol Substitution Test/Coding (DSST). The lower the score, the stronger the indication of fatigability
Self rated post-concussion symptoms | Measured at approximately one week after injury
  For assessment of self-rated symptoms The Rivermead Post-Concussion Symptoms Questionnaire (RPQ) was used. RPQ is based on a Likert scale and includes 16 items with ratings from 0 to 4. Higher score indicates more symptoms
Self rated post-concussion symptoms | Measured at approximately 4 months after injury
  For assessment of self-rated symptoms The Rivermead Post-Concussion Symptoms Questionnaire (RPQ) was used. RPQ is based on a Likert scale and includes 16 items with ratings from 0 to 4. Higher score indicates more symptoms

SECONDARY OUTCOMES:
Trait fatigability | Measured at approximately one week after injury
  The Fatigue Severity Scale (FSS) was used to measure trait fatigue. FSS consists of 9 questions and is based on a 7 point Likert scale A high score implies a higher level of fatigue.
Trait fatigability | Measured at approximately 4 months after injury
  The Fatigue Severity Scale (FSS) was used to measure trait fatigue. FSS consists of 9 questions and is based on a 7 point Likert scale A high score implies a higher level of fatigue.
Anxiety and depression | Measured at approximately one week after injury
  Hospital Anxiety and Depression (HADS) scale was used to screen for depression and anxiety, range (0-42) higher scores indicate more severe problems
Anxiety and depression | Measured at approximately 4 months after injury
  Hospital Anxiety and Depression (HADS) scale was used to screen for depression and anxiety, range (0-42) higher scores indicate more severe problems
Self-rated visual symptoms in near work | Measured at approximately one week after injury
  Convergence Insufficiency Symptom Survey (CISS) was used to assess near work-related visual symptoms. Total score is 60 and a value above 21 indicates a high level of symptoms.
Self-rated visual symptoms in near work | Measured at approximately 4 months after injury
  Convergence Insufficiency Symptom Survey (CISS) was used to assess near work-related visual symptoms. Total score is 60 and a value above 21 indicates a high level of symptoms.
Convergence | Measured at approximately one week after injury
  A visual examination performed by a licensed optometrist, using standard optometric clinical methods. Diagnosis of visual dysfunction were based on established diagnostic criteria
Convergence | Measured at approximately 4 months after injury
  A visual examination performed by a licensed optometrist, using standard optometric clinical methods. Diagnosis of visual dysfunction were based on established diagnostic criteria
Accommodation | Measured at approximately one week after injury
  A visual examination performed by a licensed optometrist, using standard optometric clinical methods. Diagnosis of visual dysfunction were based on established diagnostic criteria
Accommodation | Measured at approximately 4 months after injury
  A visual examination performed by a licensed optometrist, using standard optometric clinical methods. Diagnosis of visual dysfunction were based on established diagnostic criteria
Fusional vergence | Measured at approximately one week after injury
  A visual examination performed by a licensed optometrist, using standard optometric clinical methods. Diagnosis of visual dysfunction were based on established diagnostic criteria
Fusional vergence | Measured at approximately 4 months after injury
  A visual examination performed by a licensed optometrist, using standard optometric clinical methods. Diagnosis of visual dysfunction were based on established diagnostic criteria

CONTACTS AND LOCATIONS:
Overall Officials: Marika C Moller, PhD, Principal Investigator — Departement of Rehabilitation Medicine, Danderyd Hospital
Locations (1):
- Department of Rehabilitation Medicine, Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cassidy JD, Carroll LJ, Peloso PM, Borg J, von Holst H, Holm L, Kraus J, Coronado VG; WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. Incidence, risk factors and prevention of mild traumatic brain injury: results of the WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. J Rehabil Med. 2004 Feb;(43 Suppl):28-60. doi: 10.1080/16501960410023732. PMID 15083870
- [Background] McInnes K, Friesen CL, MacKenzie DE, Westwood DA, Boe SG. Mild Traumatic Brain Injury (mTBI) and chronic cognitive impairment: A scoping review. PLoS One. 2017 Apr 11;12(4):e0174847. doi: 10.1371/journal.pone.0174847. eCollection 2017. PMID 28399158
- [Background] Puig J, Ellis MJ, Kornelsen J, Figley TD, Figley CR, Daunis-I-Estadella P, Mutch WAC, Essig M. Magnetic Resonance Imaging Biomarkers of Brain Connectivity in Predicting Outcome after Mild Traumatic Brain Injury: A Systematic Review. J Neurotrauma. 2020 Aug 15;37(16):1761-1776. doi: 10.1089/neu.2019.6623. Epub 2020 Apr 24. PMID 32228145
- [Background] Madhavan R, Joel SE, Mullick R, Cogsil T, Niogi SN, Tsiouris AJ, Mukherjee P, Masdeu JC, Marinelli L, Shetty T. Longitudinal Resting State Functional Connectivity Predicts Clinical Outcome in Mild Traumatic Brain Injury. J Neurotrauma. 2019 Mar 1;36(5):650-660. doi: 10.1089/neu.2018.5739. Epub 2018 Oct 3. PMID 30024343
- [Background] Palacios EM, Yuh EL, Chang YS, Yue JK, Schnyer DM, Okonkwo DO, Valadka AB, Gordon WA, Maas AIR, Vassar M, Manley GT, Mukherjee P. Resting-State Functional Connectivity Alterations Associated with Six-Month Outcomes in Mild Traumatic Brain Injury. J Neurotrauma. 2017 Apr 15;34(8):1546-1557. doi: 10.1089/neu.2016.4752. Epub 2017 Jan 13. PMID 28085565
- [Background] Jones RN, Manly J, Glymour MM, Rentz DM, Jefferson AL, Stern Y. Conceptual and measurement challenges in research on cognitive reserve. J Int Neuropsychol Soc. 2011 Jul;17(4):593-601. doi: 10.1017/S1355617710001748. PMID 21411036
- [Background] Nelson ME, Jester DJ, Petkus AJ, Andel R. Cognitive Reserve, Alzheimer's Neuropathology, and Risk of Dementia: A Systematic Review and Meta-Analysis. Neuropsychol Rev. 2021 Jun;31(2):233-250. doi: 10.1007/s11065-021-09478-4. Epub 2021 Jan 8. PMID 33415533
- [Background] Sumowski JF, Rocca MA, Leavitt VM, Dackovic J, Mesaros S, Drulovic J, DeLuca J, Filippi M. Brain reserve and cognitive reserve protect against cognitive decline over 4.5 years in MS. Neurology. 2014 May 20;82(20):1776-83. doi: 10.1212/WNL.0000000000000433. Epub 2014 Apr 18. PMID 24748670
- [Background] Oldenburg C, Lundin A, Edman G, Nygren-de Boussard C, Bartfai A. Cognitive reserve and persistent post-concussion symptoms--A prospective mild traumatic brain injury (mTBI) cohort study. Brain Inj. 2016;30(2):146-55. doi: 10.3109/02699052.2015.1089598. Epub 2015 Nov 30. PMID 26618716
- [Derived] Ekdahl N, Moller MC, Deboussard CN, Stalnacke BM, Lannsjo M, Nordin LE. Investigating cognitive reserve, symptom resolution and brain connectivity in mild traumatic brain injury. BMC Neurol. 2023 Dec 20;23(1):450. doi: 10.1186/s12883-023-03509-8. PMID 38124076

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT05593172/Prot_SAP_000.pdf